CLINICAL TRIAL: NCT04059120
Title: Expression of BNDF Through Stretching as a Recovery Mechanism in Subjects With Overtraining
Brief Title: Expression of BNDF Through Stretching and Recovery
Acronym: BDNF&Exe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Colima (Other)
Responsible Party: Principal Investigator, Pedro Julian Flores Moreno, Msc, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 090128
Record Dates: First submitted 2019-03-05; First posted 2019-08-16 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Exercise
Keywords: Exercise; Overtraining; BDNF; Stretching
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The model of the physical training program to follow is. The subjects will perform a physical exercise for 12 weeks divided into three blocks of 4 periods, organized in 3 weeks of training, plus 1 rest, which simulate physical loads similar to the periods of competition used in high-performance sports. The evaluations will be made prior to the training (basal measurement) and at the end of each of the blocks during the rest period. The physical load will be organized as follows: The control group (CG) will perform muscle strength exercises with intensities of 45 to 90% of 1RM, as well as aerobic resistance with efforts of 60 to 90% of the theoretical maximum heart rate, which will be controlled with a Polar brand heart rate monitor model FT7. Like the CG, the experimental group (EG) will perform the same physical load of muscular strength and aerobic resistance in combination with specific stretching exercises
Who Masked: Participant
Masking Description: The blindness will be on the part of the subjects do not recognize the type of stretching training that is being done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The physical load will be organized as follows: The experimental group (EG) will perform muscle strength exercises with intensities of 45 to 90% of 1RM in combination with specific stretching exercises, and aerobic resistance with efforts of 60 to 90% of the theoretical maximum heart rate, which will be controlled with a Polar brand heart rate monitor model FT7.
  Interventions: Other: Experimental group whit specific stretching
- Control group (Active Comparator): The physical load will be organized as follows: The control group (CG) will perform muscle strength exercises with intensities of 45 to 90% of 1RM in combination with single or general stretching exercises, and aerobic resistance with efforts of 60 to 90% of the theoretical maximum heart rate, which will be controlled with a Polar brand heart rate monitor model FT7.
  Interventions: Other: Control group whit out specific stretching

INTERVENTIONS:
Other: Experimental group whit specific stretching — The intervention involves a reality of physical, physical, different exercise, similar to the realist of high-performance athletes. However, this is the physical load, which is reduced with specific exercises of stretching and with it the factors that determine the syndrome of overtraining
  Arms: Experimental group
Other: Control group whit out specific stretching — The intervention involves a reality of physical, physical, different exercise, similar to the realist of high-performance athletes. However, this is the physical load, which is reduced less than specific exercises of stretching and with it the factors that determine the syndrome of overtraining
  Arms: Control group

SUMMARY:
The phenomena of biological adaptation and overtraining are closely related terms, that is why in sport it is possible to identify two types of overtraining. The first of these is known as short-term overtraining, which is required as a state of peripheral fatigue induced by repeated sessions of physical activity in short periods of time that are related to mechanisms of metabolic type, is considered desirable and normal, by allowing mechanisms of adaptation to be activated depending on the nature and administration of the loads, which allow reaching higher yield quotas. The second, long-term overtraining, is characterized by a series of signs and symptoms of exhaustion and persistent fatigue that take place at the level of the central nervous system and that are produced by the imbalance between demanding physical work and recovery periods.This type of condition is also known as, general syndrome of overtraining (GSO), unexplained low performance syndrome, staleness or burnout, which is propitiated by the need to achieve maximum physical performance and the performance of physical activities in a uncontrolled that cause an interruption to the processes of biological recovery that attenuate the obtaining of the physical form wished, reason why the sportsman experiences a decrease of the physical and mental performance, manifested in a clinical picture that reflects muscular inflammation, headache, elevation sudden blood pressure, loss of functional capacity, alterations of the central nervous system (CNS), metabolic, endocrine and immune systems.

The stretching is commonly used as a method of physical rehabilitation. The actual information about how the GSO can reduce or prevent in the athlete are no cleared yet, that is the way the information regarding the relationship with the GSO, the stretching, the expression of BDNF and the effects can produce in the regenerative capacity in the over-trained subjects and their compensatory mechanisms during the different cycles of physical exercise, is null, making necessary the investigation of the effects that can produce in the decrease of factors that indicate GSO.

DETAILED DESCRIPTION:
Introduction. The phenomena of biological adaptation and overtraining are closely related terms, that is why in sport it is possible to identify two types of overtraining. The first of these is known as short-term overtraining, which is required as a state of peripheral fatigue induced by repeated sessions of physical activity in short periods of time that are related to mechanisms of metabolic type (e.g. low levels of glycogen), is considered desirable and normal, by allowing mechanisms of adaptation to be activated depending on the nature and administration of the loads, which allow reaching higher yield quotas. The second, long-term overtraining, is characterized by a series of signs and symptoms of exhaustion and persistent fatigue that take place at the level of the central nervous system and that are produced by the imbalance between demanding physical work and recovery periods.

This type of condition is also known as, general syndrome of overtraining (GSO), unexplained low performance syndrome, staleness or burnout, which is propitiated by the need to achieve maximum physical performance and the performance of physical activities in a uncontrolled that cause an interruption to the processes of biological recovery that attenuate the obtaining of the physical form wished, reason why the sportsman experiences a decrease of the physical and mental performance, manifested in a clinical picture that reflects muscular inflammation, headache, elevation sudden blood pressure, loss of functional capacity, alterations of the central nervous system (CNS), metabolic, endocrine and immune systems. The neurotrophic factor derived from the brain (BDNF) influences different types of neurons in the CNS, promoting their differentiation, growth, survival, and neuroprotection by activating the mechanisms of synaptic plasticity.

BDNF decreases when performing specific physical exercises with intensities under the interval (mixed) and high-intensity method; as those who are employed in competitive cycles. For its part, stretching is commonly used as a method of physical rehabilitation in patients with musculoskeletal injuries of various origins. Its effect reflects the restoration of motor control by interacting with the intervention and order centers that are located in different parts of the CNS that are associated with the modulation of the discharge of the motor neurons involved in the activation of the muscle spindle, which allow the reflex for the execution of the movement and the control of postures. The information regarding the relationship with the GSO, the stretching and the expression of BDNF in the regenerative capacity in those over-trained subjects and their compensatory mechanisms during the different cycles of physical exercise, is null, making necessary the investigation of the effects that can produce in the decrease of factors that indicate GSO and, consequently, build support systems for the athlete with the purpose of returning it to a level of adequate physical performance.

Problem Statement. The training cycles are configured with the purpose of achieving a greater adaptation to the physical activity that is performed. However, those closest to the competition have more intensity and physical demands. However, the achievement of maximum performance and the GSO are phenomena deeply related to the adaptability of the organism. The strategies commonly used to recover an athlete with GSO, are directed to the care of diet and rest, however, do not make clear by what methods and means it is possible to perform a restoration of regenerative processes and muscle contraction to decrease of chronic fatigue and in turn the maintenance of physical performance achieved in previous cycles.

Research question. What are the effects of a stretching training program on BDNF expression and its relationship with biochemical and physiological markers that indicate GSO?

General objective. To analyze the effects of a stretching training program on the expression of BDNF and decrease of biochemical and physiological markers that indicate GSO.

Methodology. A clinical trial, with simple blinding.

Type of sampling. Probabilistic, simple random (tombola).

Sample size. 72 subjects, 36 subjects per group, which was estimated through the equation for comparison of means.

Selection criteria. To be a university student, males from 18 to 25 years of age, to lead a moderately active or sedentary lifestyle, to sign an informed consent form, to take the physical fitness level test and to have been diagnosed as healthy in the clinical assessment.

Attention to adverse effects. These will be classified into three types, milder, will be those muscular discomforts present but tolerable, e.g. delayed muscle pain (stiffness), edema, localized fatigue, loss of mobility, loss of strength. Moderate, physical damage that interferes with physical activities, such as, first or second-degree sprain and first-degree muscle tear. Severe, those injuries and/or physical damage that incapacitates the subject to perform physical activities of any kind, such as ruptures, severe muscular, ligamentous and cartilaginous of the third degree, dislocations and fractures. If one of the two previous cases are presented, the subjects will be assisted by the sports doctor who is part of the research protocol and channeled to the corresponding family medical clinic.

Instruments. Questionnaire PAR Q & YOU used to know the state of health and habits of physical activity. The biochemical tests will be carried out with a blood sample of 5 ml using a BD Vacutainer yellow tube model 368159 with gel separator and coagulation activator, which will estimate the concentrations of creatine phosphokinase, testosterone, cortisol, and brain-derived neurotrophic factor, which will be quantified with the ELISA method. The physiological determinants will be measured with the general stretching index test (GSI), which is calculated by the sum of the stretching in sitting, standing and lying down multiplied by the body surface. The level of physical fitness will be assessed with the Tecumseh step test and the VO2max with the Astrand-Rhyming test.

Physical training program. The study subjects will perform a physical exercise for 12 weeks divided into three blocks of 4 periods, organized in 3 weeks of training, plus 1 rest, which simulate physical loads similar to the periods of competition used in high-performance sports. The evaluations will be made prior to the training (basal measurement) and at the end of each of the blocks during the rest period. The physical load will be organized as follows: The control group (CG) will perform muscle strength exercises with intensities of 45 to 90% of 1RM, as well as aerobic resistance with efforts of 60 to 90% of the theoretical maximum heart rate, which will be controlled with a Polar brand heart rate monitor model FT7. Like the CG, the experimental group (EG) will perform the same physical load of muscular strength and aerobic resistance in combination with specific stretching exercises.

Statistical analysis. Kolmogorov Smirnov test to check the normality of the data, in case of presenting a normal distribution (p <0.05) the repeated measures ANOVA test will be applied, otherwise the Kruskal Wallis test will be applied. The correlation level will be established with the Pearson or RhO Spearman test. Factorial analysis of the relationship between variables and individuals will be applied through Hj-biplot. The analysis of variables will be carried out with the SPSS v 20.0 program, establishing a level of p <0.05 as the level of statistical significance.

Ethical considerations. The protocol was approved by the Research and Ethics in Research Committee of the State Institute of Cancerology, with registration number CICC-090218-BDNFMRS-05. Financing. $ 94,764.76. At the moment there are two ELISA kits for BDNF analysis and $ 44,286.76 are being managed with the Movimiento es Salud Foundation for the purchase and/or maquila of the testosterone, cortisol and CPK samples.

ELIGIBILITY:
Inclusion Criteria:

1. Be a student of the degree in physical education and sports at the University of Colima.
2. Men with ages from 18 to 25 years.
3. Lead a moderate sedentary or active recreational lifestyle
4. Sign the act of voluntary participation in the study, with the precise knowledge of the qualifications and the procedures applied.
5. Having completed the Tecumseh test, passing the test and knowing the level of physical fitness
6. Have been diagnosed as healthy after being submitted to the clinical assessment.

Exclusion Criteria:

1. Presenting metabolic alterations such as type I or II diabetes
2. Having chronic respiratory diseases such as pulmonary, chronic obstructive disease, asthma, emphysema or cancer.
3. Having high blood pressure or arrhythmia.
4. Be under a physical training of muscular strength or aerobic resistance with high-performance direction.
5. Be under some drug treatment or drug use.

Elimination criteria

1. All subjects who wish to leave the study voluntarily
2. Those subjects who present ostiomyoarticular and skeletal injuries caused by the physical exercise performed. A medical specialist in sports medicine, a person at work, a medical care channel.
3. Subjects who present symptoms of wear or corrosion during the training received. Same that will be directed to make a break, in addition to attended and monitored by a sports doctor. From the need for more attention, they will be channeled to the familiar doctor.
4. Those who do not comply with 70% attendance to the physical training program

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Changes of the BDNF from basal levels to 1 and 3 month | Baseline, 1 month to 3 month (12 weeks)
  Measurement of serum concentration of the BDNF (pg/ml) by ELISA Method

SECONDARY OUTCOMES:
Changes in the testosterone/cortisol index from basal levels to 1 and 3 month | Baseline, 1 month to 3 month (12 weeks)
  Measurement of serum concentration of cortisol (µMol/l) and testoterone (nMol/l ) by ELISA Method
Changes of the creatine phosphokinase from basal level to 1 and 3 month | Baseline, 1 month to 3 month (12 weeks)
  Measurement of serum concentration of the creatine phosphokinase (U/L) by ELISA method

CONTACTS AND LOCATIONS:
Overall Officials: Del Río Va José Encarnación, PhD, Study Director — Universidad de Colima
Locations (1):
- Universidad de Colima, Colima, Mexico

IPD SHARING:
Plan to Share IPD: No
The volunteers data will no share whit other investigation because this project is for individual

REFERENCES:
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Background] Wilmore, JH & Costill DL Physiology of effort and sport. 2007. Paidotribo. Spain
- [Background] Meeusen R, Duclos M, Foster C, Fry A, Gleeson M, Nieman D, Raglin J, Rietjens G, Steinacker J, Urhausen A; European College of Sport Science; American College of Sports Medicine. Prevention, diagnosis, and treatment of the overtraining syndrome: joint consensus statement of the European College of Sport Science and the American College of Sports Medicine. Med Sci Sports Exerc. 2013 Jan;45(1):186-205. doi: 10.1249/MSS.0b013e318279a10a. PMID 23247672
- [Background] Wyatt, FB, Donaldson, A, & Brown, E. The overtraining syndrome: A meta-analytic review. Journal of exercise physiology. 16 (2), 12-23, 2013
- [Background] Bergado, J, Lorigados, L. Alberti, E. & Almaguer, W. Neurotrophic factor derived from the brain in brain tissue of healthy rats. Journal CENIC Biological Sciences, 2 (40), 135 - 139, 2009
- [Background] González, R, Miller, R, Martínez, R, Andrade, A & Márquez, S. Adaptation in sport and its relation to overtraining. Notebooks of sports psychology. 6 (1), 81-98, 2006.
- [Background] Huesca, JM. Analysis of the general index of flexibility. Sports medicine 71 (2): 65-69, 2004
- [Background] Mackenzie, B. 101 Performance evaluation tests. Electric Word plc. 2005
- [Result] Budgett R. Overtraining syndrome. Br J Sports Med. 1990 Dec;24(4):231-6. doi: 10.1136/bjsm.24.4.231. PMID 2097018
- [Result] Sesboue B, Guincestre JY. Muscular fatigue. Ann Readapt Med Phys. 2006 Jul;49(6):257-64, 348-54. doi: 10.1016/j.annrmp.2006.04.021. Epub 2006 Apr 27. English, French. PMID 16757054
- [Result] Kreher JB, Schwartz JB. Overtraining syndrome: a practical guide. Sports Health. 2012 Mar;4(2):128-38. doi: 10.1177/1941738111434406. PMID 23016079
- [Result] Jackson AS, Blair SN, Mahar MT, Wier LT, Ross RM, Stuteville JE. Prediction of functional aerobic capacity without exercise testing. Med Sci Sports Exerc. 1990 Dec;22(6):863-70. doi: 10.1249/00005768-199012000-00021. PMID 2287267